CLINICAL TRIAL: NCT05077982
Title: Long Term Outcomes of COVID-19 Critical Illness: Cohort Study of Adult Patients Admitted to the Intensive Care Unit at Mater Dei Hospital With COVID-19 Infection
Brief Title: The Long Term Effects of COVID on Pulmonary Function
Status: Completed | Type: Observational
Sponsor: Sciberras, Stephen M.D. (Individual)
Collaborators: Mater Dei Hospital, Malta (Other)
Responsible Party: Principal Investigator, Stephen Sciberras, Supervisor, Sciberras, Stephen M.D.
Other Study IDs: LongTermCOVID
Record Dates: First submitted 2021-08-26; First posted 2021-10-14 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Covid19; COVID-19 Pneumonia; Critical Illness; Quality of Life
Keywords: Covid19; Critical Illness
MeSH Terms: conditions — COVID-19; Critical Illness | interventions — Spirometry; Walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spirometry — Spirometry to assess lung function
Diagnostic Test: 6-minute walk — Exercise tolerance

SUMMARY:
An observational cohort study of patients discharged from the ICU following admission with COVID19 infection, looking at their medical wellbeing 6 months after discharge from the ICU.

DETAILED DESCRIPTION:
The COVID-19 epidemic has placed an unprecedented strain on medical services worldwide. Throughout 2020 and early 2021, hospitals and their critical care services have been inundated with patients suffering from critical illness due to COVID-19, some of whom developed multi-organ failure and required a prolonged ICU stay. While the medical literature is now replete with publications and research on the acute phase of illness due to COVID-19, including critical illness, there is a paucity of studies detailing the long-term outcomes following COVID-19 critical illness.

While the negative long-term physical health, mental health and quality-of-life related effects of ARDS have been well documented, there has been very little long-term COVID-19 ARDS specific outcome studies published.

This is an observational cohort study that aims to assess the long-term health outcomes of adult patients admitted to Mater Dei Hospital Intensive Care Unit with COVID-19 infection. Patients will initially be assessed at 6 months after discharge from ITU. They will be interviewed by trained researchers using validated questionnaires. These questionnaires will assess their physical health, mental health and functional status. Participants will be examined and asked to do a 6minute walk test also using validated non-invasive physical assessment tools. They will be offered pulmonary function tests to be carried out at the Pulmonary function laboratory.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Intensive Care Unit with organ failure secondary to acute COVID-19 infection and successfully discharged from Mater Dei Hospital and surviving beyond 6 months after discharge, will be offered inclusion in the study.

A positive COVID PCR result before or during the patient's admission will be necessary for inclusion in the study. Participants will be over 18 years of age, with no restriction as regards race, ethnicity or gender.

Exclusion Criteria:

* There are no exclusion criteria

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be included
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Long term general health effects of critical illness due to COVID-19 infection | at 6 months
  Observation of the effect critical illness due to COVID-19 has on a patients' health related quality of life at 6 and 12 months after discharge from the ICU
Long term general health effects of critical illness due to COVID-19 infection | at 12 months
  Observation of the effect critical illness due to COVID-19 has on a patients' health related quality of life at 6 and 12 months after discharge from the ICU

SECONDARY OUTCOMES:
Correlation between severity of COVID19 illness and QOL | at 6 months
  Observation of how different severity of critical illness secondary to COVID-19 infection correlates with medium and long-term health related quality of life outcomes.
Correlation between severity of COVID19 illness and QOL | at 12 months
  Observation of how different severity of critical illness secondary to COVID-19 infection correlates with medium and long-term health related quality of life outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Dei Hospital, Msida, Malta

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT05077982/Prot_SAP_000.pdf